CLINICAL TRIAL: NCT03234634
Title: Collateral-based reSetting of Endovascular Treatment Time Window for Stroke (CoSETS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As the guideline for the acute stroke endovascular treatment of the AHA/ASA was changed, DSMB recommended an end to the study.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2017-0511
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Patients will be dichotomized into good collateral (group 1) and poor collateral group (group 2) according to collateral status assessed on multiphase CT angiography.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: patients with good collateral (No Intervention)
- Group 2a, patient with poor collaterals (Experimental): Group 2 patients (poor collateral group) will be randomized into endovascular thrombectomy group (2a) and best medical treatment group (2b), if femoral puncture is possible between 150 minutes and 600 minutes after last seen well.
  Interventions: Procedure: endovascular thrombectomy
- Group 2b, patients with poor collaterals (No Intervention): Group 2 patients (poor collateral group) will be randomized into endovascular thrombectomy group (2a) and best medical treatment group (2b), if femoral puncture is possible between 150 minutes and 600 minutes after last seen well.

INTERVENTIONS:
Procedure: endovascular thrombectomy — Intervention description : Group 1: patients with good collateral, Group 2: patient with poor collateral
  1. Group 1 patients (good collateral group) will receive endovascular thrombectomy using stent retriever, aspiration catheter, or both, if femoral puncture is possible between 150 minutes and 600 minutes after last seen well.
  2. Group 2 patients (poor collateral group) will be randomized into endovascular thrombectomy group (2a) and best medical treatment group (2b), if femoral puncture is possible between 150 minutes and 600 minutes after last seen well.
  Other Names: best medical treatment
  Arms: Group 2a, patient with poor collaterals

SUMMARY:
This study is a prospective, partly randomized, multi-center, Phase III, controlled trial, designed to show that the onset-to-puncture time (OPT) for good functional outcome (defined by modified Rankin Scale score at 3 months, 0-2) can be set depending on collateral status based on multiphase CT angiogram. The purpose of this study is to prove that (1) for patients with poor collaterals, there will no difference in good outcome rate between endovascular treatment and best medical treatment group if onset-to-puncture time is between 150 minutes and 600 minutes, and 2) for patients wih good collaterals, the rate of good outcome is equal to or greater than 42% (10% greater than historical control) if onset-to-puncture time is between 150 minutes and 600 minutes. Patients will initially be classified into 3 arms based on both collateral status on multiphase CT angiography and whether or not receiving endovascular thrombectomy: group 1, patients with good collaterals and receiving endovascular thrombectomy, 2) group 2a, patient with poor collaterals and receiving endovascular thrombectomy, and 3) group 2b, patients with poor collaterals and not receiving endovascular thrombectomy. Patients with good collaterals will receive endovascular thrombectomy (EVT) if onset-to-puncture time is between 150 minutes and 600 minutes after last seen well time. Of the patients with poor collaterals, they will be randomized into endovascular treatment and best medical treatment group, if onset-to-puncture time is between 150 minutes and 600 minutes, (onset-to-puncture time is not possible within 150 minutes but possible within 600 minutes after last seen well). Primary endpoint is the rate of good outcome at 3 months. The number of subjects needed with statistical power of 0.8 and alpha value of 0.025 is estimated 309 patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* Age ≥ 19 years old
* Modified Rankin Scale score before qualifying stroke, 0 or 1
* Baseline National Institute of Health Stroke Scale, 5 or greater
* Baseline Alberta Stroke Program Early Computed Tomographic Sign, 6 or greater
* Documented occlusion of relevant intracranial internal carotid artery or middle cerebral artery M1 segment on multiphase CT angiogram
* Starting of endovascular treatment (femoral artery puncture) should be possible between 150 minutes and 600 minutes after last seen well time.
* Nonenhanced CT and multiphase CT angiogram should be obtained in the participating hospital
* If indicated, intravenous administration of tissue plasminogen activator should be given.

Exclusion Criteria:

* Femoral puncture is impossible
* Pregnancy or positive on serum beta-hCG test
* Known uncontrollable allergic reaction to iodized contrast media
* Intracranial cerebral artery dissection
* Suspected chronic occlusion of the relevant intracranial large artery
* In hospital stroke
* Bilateral internal carotid artery or middle cerebral artery occlusion
* Underlying severe medical or surgical disease which may affect treatment response.
* Clinical follow is impossible because of social or medical problems.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
The rate of good functional outcome defined by modified Rankin Scale score 0 - 2 | 90 days ± 14 days after enrollment
  The scale runs from 0-6, running from perfect health without symptoms to death 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

SECONDARY OUTCOMES:
modified Rankin Scale score | 90 days ± 14 days after enrollment
NIHSS score | 24 hours after enrollment
NIHSS score | 72 hours after enrollment
NIHSS score | 7 days after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Healthcare System, Severance Hospital, Seoul, Yeonsei-ro Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu I, Bang OY, Chung JW, Kim YC, Choi EH, Seo WK, Kim GM, Menon BK, Demchuk AM, Goyal M, Hill MD. Admission Diffusion-Weighted Imaging Lesion Volume in Patients With Large Vessel Occlusion Stroke and Alberta Stroke Program Early CT Score of >/=6 Points: Serial Computed Tomography-Magnetic Resonance Imaging Collateral Measurements. Stroke. 2019 Nov;50(11):3115-3120. doi: 10.1161/STROKEAHA.119.026229. Epub 2019 Sep 26. PMID 31554502